CLINICAL TRIAL: NCT02792400
Title: The Role of Glucagon in the Effects of Dipeptidyl Peptidase-4 Inhibitors and Sodium-glucose Co-transporter-2 Inhibitors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Sofie Hædersdal, MD, PhD student, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-15018701
Record Dates: First submitted 2016-06-01; First posted 2016-06-07 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2017-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin; empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- A1: GRA-placebo + MEAL + DPP4-placebo (Placebo Comparator): LY2409021 placebo + 4 hour standardised liquid mixed-meal test + linagliptin placebo
  Interventions: Drug: LY2403021 placebo; Procedure: Standardised liquid meal; Drug: Linagliptin placebo
- A2: GRA-active + MEAL + DPP4-placebo (Placebo Comparator): 300 mg LY2409021 + 4 hour standardised liquid mixed-meal test + linagliptin placebo
  Interventions: Drug: LY2403021; Procedure: Standardised liquid meal; Drug: Linagliptin placebo
- A3: GRA-placebo + MEAL + DPP4-active (Active Comparator): LY2409021 placebo + 4 hour standardised liquid mixed-meal test + 5 mg linagliptin (Trajenta)
  Interventions: Drug: LY2403021 placebo; Procedure: Standardised liquid meal; Drug: Linagliptin
- A4: GRA-active + MEAL + DPP4-active (Active Comparator): 300 mg LY2409021 + 4 hour standardised liquid mixed-meal test + 5 mg linagliptin (Trajenta)
  Interventions: Drug: LY2403021; Procedure: Standardised liquid meal; Drug: Linagliptin
- B1: GRA-placebo + MEAL + SGLT2-placebo (Placebo Comparator): LY2409021 placebo + 4 hour standardised liquid mixed-meal test + empagliflozin placebo
  Interventions: Drug: LY2403021 placebo; Procedure: Standardised liquid meal; Drug: Empagliflozin placebo
- B2: GRA-active + MEAL + SGLT2-placebo (Placebo Comparator): 300 mg LY2409021 + 4 hour standardised liquid mixed-meal test + empagliflozin placebo
  Interventions: Drug: LY2403021; Procedure: Standardised liquid meal; Drug: Empagliflozin placebo
- B3: GRA-placebo + MEAL + SGLT2-active (Active Comparator): LY2409021 placebo + 4 hour standardised liquid mixed-meal test + 25 mg empagliflozin (Jardiance)
  Interventions: Drug: LY2403021 placebo; Procedure: Standardised liquid meal; Drug: Empagliflozin
- B4: GRA-active + MEAL + SGLT2-active (Active Comparator): 300 mg LY2409021 + 4 hour standardised liquid mixed-meal test + 25 mg empagliflozin (Jardiance)
  Interventions: Drug: LY2403021; Procedure: Standardised liquid meal; Drug: Empagliflozin

INTERVENTIONS:
Drug: LY2403021 — Glucagon receptor antagonist
  Arms: A2: GRA-active + MEAL + DPP4-placebo; A4: GRA-active + MEAL + DPP4-active; B2: GRA-active + MEAL + SGLT2-placebo; B4: GRA-active + MEAL + SGLT2-active
Drug: LY2403021 placebo
  Arms: A1: GRA-placebo + MEAL + DPP4-placebo; A3: GRA-placebo + MEAL + DPP4-active; B1: GRA-placebo + MEAL + SGLT2-placebo; B3: GRA-placebo + MEAL + SGLT2-active
Procedure: Standardised liquid meal
Drug: Linagliptin — DPP-4-inhibitor
  Other Names: Trajenta
  Arms: A3: GRA-placebo + MEAL + DPP4-active; A4: GRA-active + MEAL + DPP4-active
Drug: Linagliptin placebo
  Arms: A1: GRA-placebo + MEAL + DPP4-placebo; A2: GRA-active + MEAL + DPP4-placebo
Drug: Empagliflozin — SGLT2-inhibitor
  Other Names: Jardiance
  Arms: B3: GRA-placebo + MEAL + SGLT2-active; B4: GRA-active + MEAL + SGLT2-active
Drug: Empagliflozin placebo
  Arms: B1: GRA-placebo + MEAL + SGLT2-placebo; B2: GRA-active + MEAL + SGLT2-placebo

SUMMARY:
In normal physiology, glucagon from pancreatic alpha cells plays an important role in maintaining glucose homeostasis via its regulatory effect on hepatic glucose production. Patients with type 2 diabetes exhibit elevated plasma glucagon levels in the fasting state, and in response to ingestion of glucose or a mixed meal.glucagon, glucagon concentrations fail to decrease appropriately and may even increase. This diabetic hyperglucagonaemia may therefore contribute importantly to the hyperglycaemia of the patients.

Several glucose-lowering treatment modalities have been shown to affect glucagon levels in patients with type 2 diabetes, but the role of glucagon in the glucose-lowering effects of these treatment modalities has been difficult to discern. By using a glucagon receptor antagonist (GRA) the investigators will exploit glucagon receptor antagonism to delineate the role of glucagon during treatment with sodium-glucose co-transporter 2 (SGLT2) inhibitors and dipeptidyl peptidase 4 (DPP-4) inhibitors, which have been shown to increase and decrease plasma glucagon levels, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Caucasians above 30 years of age with diet or metformin treated type 2 diabetes for at least 3 months (diagnosed according to the criteria of the World Health Organization)
* Normal haemoglobin
* Informed consent

Exclusion Criteria:

* Inflammatory bowel disease
* Intestinal resections
* Nephropathy (serum creatinine above normal range and/or albuminuria)
* Liver disease (serum alanine aminotransferase (ALAT) and/or serum aspartate aminotransferase (ASAT) >2×normal values)
* Treatment with medicine that cannot be paused for 12 hours
* Pregnancy and/or breastfeeding
* Family history of pancreatic islet tumours
* Age above 75 years
* Treatment with loop-diuretics (applies only to arms with empagliflozin or empagliflozin placebo)
* Chronic heart failure

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05; Primary Completion 2016-08 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Difference in postprandial glucose excursions (linagliptin) | Area under the curve (AUC) time frame: 0, 5, 10, 15, 20, 25, 30, 40, 50, 60, 70, 80, 90, 105, 120, 150, 180, 210, 240 minutes. Comparison between experimental days with linagliptin (A1, A2, A3, A4)
  Difference in postprandial glucose excursions (measured as incremental (baseline substracted) area under the curve (AUC) values).
Difference in postprandial glucose excursions | Area under the curve (AUC) time frame: 0, 5, 10, 15, 20, 25, 30, 40, 50, 60, 70, 80, 90, 105, 120, 150, 180, 210, 240 minutes. Comparison between experimental days with empagliflozin (B1, B2, B3, B4)
  Difference in postprandial glucose excursions (measured as incremental (baseline substracted) area under the curve

SECONDARY OUTCOMES:
Endogenous glucose production | Plasma concentration of 6,6^2 H2-glucose and U-13C^6-glucose at times: 0,10, 20, 30, 50, 60, 70, 90, 105, 120, 150, 240 minutes.
  Glucose rate of appearance will be calculated by the non-steady state equation using double tracer technique.
Lipolysis | Plasma concentration of 1,1,2,3,3-^2-H5 - glycerol measured at times: 0,10, 20, 30, 50, 60, 70, 90, 105, 120, 150, 240 minutes.
  Glycerol disappearance will be calculated by the non-steady state equation using double tracer technique.
Serum/plasma concentrations of insulin, C-peptide, glucagon, GIP and GLP-1. | : 0,10, 20, 30, 50, 60, 70, 90, 105, 120, 150, 240 minutes
Appetite | VAS scales will be handed out at time 0, 30, 60, 90, 120, 150, 180 and 240 minutes.
  Appetite will be evaluated with a visual analogue scale (VAS).
Energy intake (kcal/kJ) | At time 240 to 270, the participants will eat an ad libitum meal.
  At the end of the standardised liquid meal test, food intake will be examined with an ad libitum meal. The weight of the food will be measured in grams and calculated to the energy intake in kcal/kJ
Changes in blood pressure (mmHg) | Measured at time 0 and time 210 minutes.
Changes in pulse rate (beat per minute) | Measured at time 0 and at time 210 minutes.
Differences in gastric emptying | -30,-15, 0, 10, 20, 30, 50, 70, 90, 105, 120, 150, 240 minutes
  Measurement of p-paracetamol. Measurement of time to peak and incremental area under the curve (iAUC)
Free fatty acids | -30,-15, 0, 10, 20, 30, 50, 70, 90, 105, 120, 150, 240 minutes
  Serum values of free fatty acids
Plasma Fibroblast growth factor-21 | -30,-15, 0, 10, 20, 30, 50, 70, 90, 105, 120, 150, 240 minutes
Resting energy expenditure | -60 to -50 and 35 to 45
  Resting energy expenditure evaluated by 10 minutes of indirect calorimetry.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Diabetes Research, Gentofte Hospital, Copenhagen University, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Haedersdal S, Lund A, Nielsen-Hannerup E, Maagensen H, van Hall G, Holst JJ, Knop FK, Vilsboll T. The Role of Glucagon in the Acute Therapeutic Effects of SGLT2 Inhibition. Diabetes. 2020 Dec;69(12):2619-2629. doi: 10.2337/db20-0369. Epub 2020 Oct 1. PMID 33004472
- [Derived] Cox AR, Chernis N, Bader DA, Saha PK, Masschelin PM, Felix JB, Sharp R, Lian Z, Putluri V, Rajapakshe K, Kim KH, Villareal DT, Armamento-Villareal R, Wu H, Coarfa C, Putluri N, Hartig SM. STAT1 Dissociates Adipose Tissue Inflammation From Insulin Sensitivity in Obesity. Diabetes. 2020 Dec;69(12):2630-2641. doi: 10.2337/db20-0384. Epub 2020 Sep 29. PMID 32994273